CLINICAL TRIAL: NCT01149213
Title: An Open-label, Follow-up Study on Remitted Patients With Major Depressive Disorder Using Transcranial Direct Current Stimulation
Brief Title: Follow-up Study of Transcranial Direct Current Stimulation to Treat Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Brunoni, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USP-HU-003
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; follow-up; relapse; remission; transcranial direct current stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental): In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp (which is located on the intersection of the sagittal and median curves). The device will deliver a charge of 2mA for 30 minutes.
  The patient will receive tDCS every other week during the first three months, then once a month during the next three months.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS will be applied at 2mA/30 minutes, every other week during the first three months than once a month during the next three months.

SUMMARY:
The investigators purpose is to follow remitted patients from their previous study using transcranial direct current stimulation (tDCS); as to verify whether this treatment prevents relapse.

DETAILED DESCRIPTION:
Our first ongoing study (Efficacy Study of Transcranial Direct Current Stimulation (tDCS) to Treat Major Depressive Disorder) addresses whether tDCS is an effective treatment for depression treatment. The purpose of the present study is to determine whether tDCS is also an effective strategy for sustaining remission.

We will enroll patients who presented remission using tDCS from our previous study and offer them to tDCS every other week for three months, than once a month for another three months. We will address whether tDCS prevents relapse by assessing depression scores once a month, using a time-to-event analysis.

The importance of the present study is to determine whether tDCS is able to sustain remission during long-term follow-up of depressed patients.

ELIGIBILITY:
Inclusion criteria:

Patients from previous studies (ID:USP-HU-001 and ID:USP-HU-002) who:

* received tDCS and responded.
* received tDCS + sertraline and responded.
* received sertraline or placebo and did not respond, and thereafter received tDCS during the cross-over phase and responded.

Exclusion criteria:

Patients from previous studies who:

* received tDCS and did not respond.
* received tDCS + sertraline and did not respond.
* received sertraline or placebo and responded.
* did not respond during the crossover phase.
* do not wish to participate in the present study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Relapse from depression | Week 4
  Once a month, we will address whether the patient has relapsed.
  Relapse criteria:
  * 2 consecutive MADRS scores > 12 or
  * any MADRS scores > 15 or
  * suicidal attempt or
  * severe suicidal ideation or
  * psychiatric hospitalization
Relapse from depression | Week 8
  Same as above.
Relapse from depression | Week 12
  Same as above.
Relapse from depression | Week 16
  Same as above.
Relapse from depression | Week 20
  Same as above.
Relapse from depression | Week 24
  Same as above.

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil